CLINICAL TRIAL: NCT02364700
Title: Hand Training Utilizing an Electromyography-triggered Hand Robot for Individuals After Chronic Stroke
Brief Title: Portable EMG-triggered Hand Robot for Individuals After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab-Robotics Company Limited (Industry)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1409015458
Record Dates: First submitted 2015-02-05; First posted 2015-02-18 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Stroke
Keywords: stroke, robotics, hand rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- interventional group (Experimental): This is a single group, interventional pilot study. All participants will receive 6-week hand training on the HOH device.
  Interventions: Device: Hand of Hope (HOH)

INTERVENTIONS:
Device: Hand of Hope (HOH) — Subjects will receive arm training 3x/week for 6 weeks, each session is anticipated to last approximately 60 minutes. Sessions will be scheduled for Monday, Wednesday, and Friday whenever possible to provide a rest period between sessions. Each session will consist of the following:
  * warm up-passive stretch of hand in flexion and extension (5 minutes);
  * setting the EMG threshold parameters for the device;
  * active practicing of opening the hand (Desperate Bee, Hungry Bird, Sun Archer games; 10 min)
  * active practice of closing then hand (UFO Catcher game; 10 min)
  * open and closing the hand (Ball and Basket game; 10 min)
  * open and closing the hand while incorporating reach ( for subjects with adequate ability to reach with shoulder/elbow; 10 min)
  * cool down-passive stretch of hand in flexion and extension (5 minutes)

SUMMARY:
This is an interventional pilot study investigating the feasibility of using the hand of hope (HOH) device for individuals with decreased hand function after stroke.

DETAILED DESCRIPTION:
The HOH will be used to provide hand training for patients with decreased hand ability after stroke. The HOH is a light-weight, non-invasive, portable hand robot that provides physical assistance when a patient activates the muscles that open and close the hand. The HOH works by detecting surface EMG muscle activity and therefore requires active participation from the patient throughout the session. Video games linked to the HOH device are specifically designed to work on opening and closing the hand facilitating mass practice and high repetition needed for improving strength and range of motion of muscles.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of stroke > 6 months ago
2. Presence of some active range of motion (AROM) in the affected hand, measured by a score of at least 1 on the Box and Block test.
3. Intact sensation in the affected hand
4. Full passive range of motion (PROM) in mass flexion and extension of the hand
5. MAS score < 3 for finger flexors and intrinsics
6. MAS score < 3 for finger extensors
7. Visual tracking is intact in all directions
8. Patient must be otherwise medically stable in the opinion of the principal investigator

Exclusion Criteria:

1. Patient is receiving active occupational or physical therapy for the affected arm
2. Patient has joint contractures that prevent proper fit into the HOH device
3. Patient has other concurrent neurological or orthopedic diagnoses that affect motor ability of the arm such as Parkinson's or Multiple Sclerosis, or arthritis
4. It has been less than 3 months since last botulinum toxin injection in the affected arm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NewYork Presbyterian Hospital-Weill Cornell Medical Center, New York, New York, United States

REFERENCES:
- [Background] O'Dell MW, Lin CC, Harrison V. Stroke rehabilitation: strategies to enhance motor recovery. Annu Rev Med. 2009;60:55-68. doi: 10.1146/annurev.med.60.042707.104248. PMID 18928333
- [Background] Tong KY, Ho SK, Pang PK, Hu XL, Tam WK, Fung KL, Wei XJ, Chen PN, Chen M. An intention driven hand functions task training robotic system. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:3406-9. doi: 10.1109/IEMBS.2010.5627930. PMID 21097247
- [Result] Ho NS, Tong KY, Hu XL, Fung KL, Wei XJ, Rong W, Susanto EA. An EMG-driven exoskeleton hand robotic training device on chronic stroke subjects: task training system for stroke rehabilitation. IEEE Int Conf Rehabil Robot. 2011;2011:5975340. doi: 10.1109/ICORR.2011.5975340. PMID 22275545
- [Result] Hu XL, Tong KY, Wei XJ, Rong W, Susanto EA, Ho SK. The effects of post-stroke upper-limb training with an electromyography (EMG)-driven hand robot. J Electromyogr Kinesiol. 2013 Oct;23(5):1065-74. doi: 10.1016/j.jelekin.2013.07.007. Epub 2013 Aug 7. PMID 23932795
- [Result] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional Group: This is a single group, interventional pilot study. Participants will received 6-week hand training on the HOH device.
  Subjects will receive arm training 3x/week for 6 weeks
Period: Overall Study
Arm/Group | Interventional Group
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Interventional Group: This is a single group, interventional pilot study. All participants will receive 6-week hand training on the HOH device. Subjects will receive arm training 3x/week for 6 weeks.
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Box and Blocks [Mean (Standard Deviation); unit: number of blocks] — This is a performance-based assessment of unilateral gross manual dexterity of the upper extremity in adults after stroke. The total score is the number of 2.5cc blocks successfully transferred with the affected hand from one box to another in one minute.
  number of blocks | 5.67 (10.36)
Arm Motor Ability Test (AMAT) [Mean (Standard Deviation); unit: units on a scale] — Performance-based measure to assess ability of participant to perform everyday functional upper extremity tasks unilaterally or bilaterally. Scoring is based on a 0-5 ordinal scale, with 0 being no ability and 5 being normal arm ability (highest score). It is comprised on 10 functional tasks. The total score is the average of scores on individual task items combined.
  units on a scale | 2.13 (.50)
Fugl-Meyer Assessment (FMA) [Mean (Standard Deviation); unit: units on a scale] — The FMA is a widely-used performance-based measure of impairment for nine upper extremity movements. It examines flexor and extensor synergy patterns, movements out of synergy patterns, wrist and hand movements, as well as strength and coordination of fine motor movements. Scores range from 0-66, with 66 being the highest score possible. For this study, the three reflex items were omitted from the final score because it is considered a separate construct from motor impairment making the maximum score 60.
  units on a scale | 20.75 (7.90)
Stroke Upper Limb Capacity Scale (SULCS) [Mean (Standard Deviation); unit: units on a scale] — The SULCS was developed to measure the capacity of the affected upper limb after stroke. Each of the 10 items arranged in a hierarchical order is assigned a score of 0 (unable to complete) or 1 (able to complete the task) with a maximum score of 10.
  units on a scale | 5.33 (2.15)
Stroke Impact Scale-Hand Subscale [Mean (Standard Deviation); unit: units on a scale] — The Stroke Impact Scale is a stroke-specific questionnaire evaluating quality of life in stroke survivors over eight domains. Each domain is scored independently on an ordinal scale ranging from 0 to a maximum of 5. Only the Hand sub-score (SIS-H) was used in this study. Scores for each domain are transformed and range from 0-100.
  Formula for scoring domains:
  Transformed Scale = [(Actual raw score - lowest possible raw score) / Possible raw score] * 100
  units on a scale | 11.50 (4.91)
Dynamometry [Mean (Standard Deviation); unit: kilograms] — Dynamometer is a valid and reliable assessment of grip strength (impairment) measured in kilograms.
  kilograms | 7.96 (6.24)

OUTCOME MEASURES:

1. Primary Outcome: Fugl-Meyer Assessment of Upper Extremity (FMA)
Description: The FMA is a performance based evaluation of upper limb impairment of the affected arm after stroke. Scoring is based on an ordinal scale of 0 (no movement) to 2 (normal movement). Scoring is based on sum of 30 items, ranging from 0-60.
Time Frame: baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
units on a scale | 22.50 (9.47)
Statistical Analysis 1: Comparison: Interventional Group; Test type: Equivalence — Group means from baseline to discharge were compared to determine if 6-week and training on the Hand of Hope device elicited changes in outcome measures; p < .05, Friedman Test

2. Primary Outcome: Arm Motor Ability Test (AMAT)
Description: The AMAT is performance based measure of functional ability of the affected arm and hand in unilateral and bilateral everyday tasks. It is comprised of 10 functional tasks such as cutting meat with a knife and fork, donning a t-shirt, and phone use with a score ranging from 0 to a maximum of 5 for each item. The total score is the mean score for all individual item scores.
Time Frame: Baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
units on a scale | 2.35 (0.58)

3. Primary Outcome: Box and Blocks
Description: The Box and Blocks is a performance-based functional assessment of hand dexterity ( gross grasp and release). The total score is the number of 2.5cc blocks successfully transferred from one box to another with the affected hand in one minute.
Time Frame: Baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: totally number of blocks transferred
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
totally number of blocks transferred | 6.08 (10)

4. Secondary Outcome: Stroke Upper Limb Capacity Scale (SULCS)
Description: The SULCs is a performance based measure of upper limb capacity after stroke. Each of the 10 items are administered in a hierarchical order and assigned a score of 0 (unable to complete) or 1 (able to complete the task) with a maximum score of 10.
Time Frame: Baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
units on a scale | 5.17 (2.17)

5. Secondary Outcome: Hand Dynamometry
Description: A dynamometer measures grip strength in kilograms
Time Frame: baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
kilograms | 8.23 (6.18)

6. Secondary Outcome: Stroke Impact Scale --Hand Sub Scale (SIS-H)
Description: The Stroke Impact Scale is a stroke-specific questionnaire evaluating quality of life in stroke survivors over eight domains. Each domain is scored independently on an ordinal scale ranging from 0 (minimum) bto a maximum of 5. Only the Hand sub-score was used in this study. Scores for each domain are transformed and range from 0-100.
  Formula for scoring domains:
  Transformed Scale = [(Actual raw score - lowest possible raw score) / Possible raw score] * 100
Time Frame: baseline to 6 weeks (discharge)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interventional Group
Number analyzed (Participants) | 12
units on a scale | 13.33 (5.48)

ADVERSE EVENTS:
Arm/Group | Interventional Group
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 7/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Group (N=12)
mild skin rubbing (Skin and subcutaneous tissue disorders) | 7 (7) — 7 subjects reported mild skin rubbing/pinching on proximal interphalangeal joint related to changes in fit of the device during training. Symptoms resolved with positional re-adjustment and/or added padding to hand (padding on finger joint or glove)
fatigue (cognitive) (General disorders) | 3 (3) — 3 participants experienced feeling tired (attention) toward end of hand training sessions. Short rest breaks used to alleviate symptoms. Did not interfere with participation
shoulder fatigue (Musculoskeletal and connective tissue disorders) | 6 (6) — 6 subjects reported muscle fatigue at shoulder during training as a results of active use. Did not interfere with study participation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No